CLINICAL TRIAL: NCT01317719
Title: Prospective Biceps Study
Status: Completed | Type: Observational
Sponsor: West Penn Allegheny Health System (Other)
Responsible Party: Principal Investigator, Carmen Latona, PI, West Penn Allegheny Health System
Other Study IDs: RC-5159
Record Dates: First submitted 2011-03-16; First posted 2011-03-17 (Estimated); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Biceps Tendon Rupture
Keywords: Rupture of Distal Bicep Tendon

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Distal Biceps Ruptures
  Interventions: Procedure: Distal Biceps Re-Insertion Surgery

INTERVENTIONS:
Procedure: Distal Biceps Re-Insertion Surgery — Surgical Repair of the Distal Biceps Tendon

SUMMARY:
The primary goal of this study is to determine if surgical repair of the distal biceps fully restores the supination strength of the forearm. Secondarily, the investigators want to examine the insertion site location of the tendon and determine if it correlates with the patients' functional outcome as determined by Disabilities of the Arm, Shoulder, and Hand (DASH), Visual Analog Pain Scale (VAPS), and isometric supination torque testing.

ELIGIBILITY:
Inclusion Criteria:

* primary distal biceps repair with endobutton

Exclusion Criteria:

* any ipsilateral wrist, forearm, or elbow condition
* any contraindication to having an MRI

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have received primary distal biceps repair by Dr. Schmidt
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2011-01-14 (Actual); Primary Completion 2013-12-30 (Actual); Study Completion 2013-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher C Schmidt, MD, Principal Investigator — WPAHS
Locations (1):
- Allegheny Imaging of McCandless, Pittsburgh, Pennsylvania, United States